CLINICAL TRIAL: NCT06356831
Title: National Registry of Surgical Treatment and Percutaneous Cryoablation of Parietal Endometriosis
Acronym: Endomercyo
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: Endomecryo
Record Dates: First submitted 2024-03-19; First posted 2024-04-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Cryotherapy Effect; Surgical; Radiology
Keywords: endometriosis; Cryo ablation; Surgical operation; radiology
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
National multicentric registry of a cohort of patient with suffering parietal endometriosis, carried out by a multidisciplinary radiosurgery team

DETAILED DESCRIPTION:
Patient who suffering of parietal endometriosis treat by cryoablation or chirurgical will be recorded in national registry. the patient will be follow during 3 years after treatement.

ELIGIBILITY:
Inclusion Criteria:

* Presence of parietal endometriosis: with suggestive clinical and imaging criteria (MRI and ultrasound)
* Symptomatic parietal endometriosis (VAS > 3 OR bothersome bleeding OR reported impact on quality of life)

Exclusion Criteria:

* Endometriosis not affecting the anterior wall of the abdomen (as deep pelvic muscle: ilio-psoas, obturators, perineal, ischio-anal fossa)
* Minor patient (< 18 years)
* Pregnant patient at any trimester
* Patient with hemostasis disorders (constitutional or acquired)
* Patient with systemic infection or localized scar infection upon inclusion.
* Patient with contraindications to MRI
* Female patient with a planned medical or surgical procedure for the duration of the study that may interfere with the proper conduct of the study.
* Patient unable to understand the information provided
* Patient who is not affiliated to the social security system
* Patient under curatorship or tutorship
* Patient with a nodule of primary or secondary malignant tumor origin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with endomecriosis at least 18 years of age who will be oer are treate by cryo ablation or surgical treatement
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
creation of a national registry for the removal of nodules by cryoablation or surgery for parietal endometriosis | at inclusion
  number of Endometriosis 's patient treat by cryoablation or surgical

SECONDARY OUTCOMES:
Characterize the epidemiology of parietal endometriosis nodules | at 1 month, 6month 1year 2 years and 3 years after treatmeant
  average of parietal endometriosis nodules
Characterize the epidemiology of parietal endometriosis nodules | at inclusion
  average of parietal endometriosis nodules
To assess the impact of hormone treatment on parietal endometriosis | at 1 month, 6month 1year 2 years and 3 years after treatmeant
  number of hormone treatment on parietal endometriosis
Assess the demographic distribution of parietal endometriosis | At inclusion
  compare the size of of endometriosis nodules pre- and post-treatment
Evaluate pre- and post-treatment imaging characteristics of parietal endometriosis | through study completion average 3 years
  compare the size of of endometriosis nodules pre- and post-treatment
Evaluate the aesthetic impact of the treatments | at 1 month after treatmeant
  number of complication
Assess the complication rate between the two groups | at 1 month, 6month 1year 2 years and 3 years after treatmeant
  number of complication between the two groups
Assess the Severity of Complications according to Society (SIR) of Interventional Radiology or Cardiovascular and Interventional Radiological Society of Europe ( CIRSE) for Radiologists | at inclusion
  average of Complications according to SIR or CIRSE for Radiologists
Assess the Severity of Complications according to Clavien Dindo for the surgeon | at inclusion
  average of Complications according to Clavien Dindo for the surgeon
Assess the recidivism rate at 3 years | at 3 years
  number of recidivism at 3 years
Assess the quality of life between the two groups with PGIC-7 questionnaire | at inclusion,1 month, 6 months 1year 2 years and 3 years after treatmeant
  average Patient Global Impression of Change PGIC-7 score : PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Assess the quality of life between the two groups with asses EHP-5 questionnaire | at inclusion,1 month, 6 months 1year 2 years and 3 years after treatmeant
  average EHP-5 score ( Endometriosis Health Profil -5). Each item is rated on a four-point scale (never = 0, rarely = 1, sometimes = 2, often = 3, always = 4 and not relevant if not applicable). Scores on the EHP-5 core and modular questionnaire then are transformed on a scale of 0 (indicating best possible health status) to 100 (indicating worst possible health status)
Assess the quality of life between the two groups with asses VAS questionnaire | at inclusion,1 month, 6 months 1year 2 years and 3 years after treatmeant
  average VAS score ( Analog Visual Scale) : VAS measures pain intensity on a scale from 0 to 10 (or sometimes from 0 to 100)
Evaluate signal and morphology changes on imaging MRI of parietal endometriosis nodules after cryoablation treatment | at inclusion,1 month, 6 months 1year 2 years and 3 years after treatmeant
  average of size of endometriosis nodules after cryoablation treatment
Evaluate signal and morphology changes on ultrasound imaging of parietal endometriosis nodules after cryoablation treatment | at inclusion,1 month, 6 months 1year 2 years and 3 years after treatmeant
  average of size endometriosis nodules after cryoablation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Léo RAZAKAMAMANTSOA, Principal Investigator — CHIC
Locations (18):
- France (18):
  - CHU bordeaux, Bordeau
  - Clinique Tivoli, Bordeaux
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHI Creteil, Créteil
  - Lyon Hôpital La Croix Rousse, Lyon
  - Lyon Hôpital Sud, Lyon
  - Lyon Louis Pradel, Lyon
  - APHM-Hôpital Nord, Marseille
  - APHP-Hôpital la Conception La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nime, Nîmes
  - AP-HP - Tenon, Paris
  - AP-HP Hôpital Européen Georges Pompidou, Paris
  - APHP Cochin-Port Royal, Paris
  - APHP-La Pitié, Paris
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CH Valencienne, Valenciennes